CLINICAL TRIAL: NCT01890642
Title: Use Of The Needle Free Jet-Injection System With Buffered Lidocaine (J-Tip) For The Treatment Of Pain During Venipuncture For Blood Draws In Young Children
Brief Title: The Use of Jet Injection Lidocaine for Blood Draws in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 443133-1
Record Dates: First submitted 2013-06-24; First posted 2013-07-02 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Pain; Children; Venipuncture; J tip; Lidocaine; video observation
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sucrose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- J tip Noise (Sham Comparator): This group will have a J tip deployed without medication to create the noise that the device makes. They will also receive Pain Ease spray if > age 1 yr or sucrose if < 1 yr
  Interventions: Device: J tip; Other: Pain Ease Spray; Other: Sucrose
- Pain Ease (Other): This group will receive Pain Ease Spray only if > 1 yr or sucrose only if child < 1 yr
  Interventions: Other: Pain Ease Spray; Other: Sucrose
- J tip (Experimental): This group will receive 1% buffered lidocaine via Jet Injection. They will receive placebo cooling spray (normal saline spray) to maintain blinding if > 1 yr and will receive sucrose is < 1 yr
  Interventions: Device: J tip; Drug: 1% buffered lidocaine; Other: placebo cooling spray (normal saline spray); Other: Sucrose

INTERVENTIONS:
Device: J tip — This is a Jet Injection system which for our study will be loaded with 1% buffered lidocaine
  Arms: J tip; J tip Noise
Other: Pain Ease Spray — Cold Spray used to anesthetize the skin
  Other Names: Cooling Spray
  Arms: J tip Noise; Pain Ease
Drug: 1% buffered lidocaine — Lidocaine placed using Jet Injection
  Other Names: Lidocaine
  Arms: J tip
Other: placebo cooling spray (normal saline spray) — Normal Saline Sprayed as placebo for Pain Ease spray
  Other Names: Normal Saline Spray
  Arms: J tip
Other: Sucrose — Oral Sucrose used for children < 1 year
  Other Names: Sweetease

SUMMARY:
This study looks at the use of Jet Injection Lidocaine (J tip) for pain during blood draws in children ages 6 and younger. The investigators will use video observation of patients to asses their pain during lab draws using either 1) Jet Injected lidocaine ( J tip) 2) Pain Ease spray 3) Pain Ease spray plus the J tip noise.

DETAILED DESCRIPTION:
No change since last report.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months-6 years seen in the Children's Hospital of Wisconsin outpatient laboratory that have an order for venipuncture for a blood draw

Exclusion Criteria:

* Previous adverse reaction to lidocaine or Pain Ease spray
* Pre-existing skin lesion at site of blood draw
* Needle stick for IV insertion or lab draw that has already occurred at current hospital visit
* Patients who are physically unable to move their arms or legs
* Patients who are unable to cry
* Patients with connective tissue disorders that predispose to easy bruising
* Patients with bleeding disorders

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maren Lunoe, MD, Principal Investigator — Medical College of Wisconsin; Amy Drendel, DO, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Lunoe MM, Bolin AE, Drendel AL. An Evaluation of High Preprocedural Anxiety and Venipuncture Pain Experienced by Young Children. Pediatr Emerg Care. 2021 Oct 1;37(10):e621-e624. doi: 10.1097/PEC.0000000000002424. PMID 34591812

RESULTS

PARTICIPANT FLOW:
Groups:
- J Tip Noise: This group will have a J tip deployed without medication to create the noise that the device makes. They will also receive Pain Ease spray
  J tip: This is a Jet Injection system which for our study will be loaded with 1% buffered lidocaine
  Pain Ease Spray: Cold Spray used to anesthetize the skin
- Pain Ease: This group will receive Pain Ease Spray
  Pain Ease Spray: Cold Spray used to anesthetize the skin
- J Tip: This group will receive 1% buffered lidocaine via Jet Injection. They will receive placebo cooling spray (normal saline spray) to maintain blinding
  J tip: This is a Jet Injection system which for our study will be loaded with 1% buffered lidocaine
  1% buffered lidocaine: Lidocaine placed using Jet Injection
  placebo cooling spray (normal saline spray): Normal Saline Sprayed as placebo for Pain Ease spray
Period: Overall Study
Arm/Group | J Tip Noise | Pain Ease | J Tip
Started | 56 | 53 | 96
Completed | 56 | 53 | 96
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | J Tip Noise | Pain Ease | J Tip | Total
Number analyzed (Participants) | 56 | 53 | 96 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 53 | 96 | 205
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.6) | 2.9 (1.7) | 3.3 (1.9) | 3.2 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 42 | 83
  Male | 31 | 37 | 54 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 21 | 38
  White | 34 | 31 | 45 | 110
  More than one race | 6 | 3 | 16 | 25
  Unknown or Not Reported | 8 | 9 | 12 | 29
Region of Enrollment [Number; unit: participants]
  United States | 56 | 53 | 96 | 205
Previous Venipuncture [Number; unit: participants] — Reported Previous Venipuncture Experience. 3 parents stated they did not know if their child had previous venipuncture, accounting for the difference between the number enrolled in the study and the number on which this variable was collected.
  participants | 55 | 51 | 96 | 202

OUTCOME MEASURES:

1. Secondary Outcome: Pain Score
Description: Pain score as assessed by video reviewers. The FLACC (Face, legs, activity, cry and consolability) Scale, ranging from 0 (no pain) to 10 (worst pain), was used to assess pain.
Time Frame: At venipuncture (3 minutes)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | J Tip Noise | Pain Ease | J Tip
Number analyzed (Participants) | 56 | 53 | 96
units on a scale | 5.75 [2.75 to 9] | 8 [3.5 to 10] | 5.25 [1.5 to 8.25]
Statistical Analysis 1: Comparison: J Tip Noise vs Pain Ease vs J Tip; Test type: Superiority or Other; p = 0.01, Kruskal-Wallis

2. Secondary Outcome: Fist Attempt Success
Description: Proportion of patients where blood draw was successful on first attempt
Time Frame: up to 3 minutes
Measure: Number; unit: participants
Arm/Group | J Tip Noise | Pain Ease | J Tip
Number analyzed (Participants) | 56 | 53 | 96
participants | 52 | 48 | 86
Statistical Analysis 1: Comparison: J Tip Noise vs Pain Ease vs J Tip; Test type: Superiority or Other; p = 0.80, Kruskal-Wallis

3. Secondary Outcome: Change in Pain Score From Baseline
Description: Pain score assessed by video reviewer before intervention (0 minute) and at venipuncture (3 minutes). The score at baseline was subtracted from the score at venipuncture to give a number indicating the change in pain scores.
  The FLACC (Face, legs, activity, cry and consolability) Scale, ranging from 0 (no pain) to 10 (worst pain), was used to assess pain.
Time Frame: 3 min
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | J Tip Noise | Pain Ease | J Tip
Number analyzed (Participants) | 56 | 53 | 96
units on a scale | 2.32 (0.48) | 3.7 (0.49) | 1.58 (0.31)
Statistical Analysis 1: Comparison: J Tip Noise vs Pain Ease vs J Tip; Test type: Superiority or Other; p = 0.004, Kruskal-Wallis

4. Primary Outcome: Change in Pain Score on FLACC Scale From Device Deployment to Venipuncture
Description: Pain score assessed by video reviewer at J-tip, J-tip noise or researcher approach (1 minute) and at venipuncture (3 minutes). The score at J-tip noise/researcher approach was subtracted from the score at venipuncture to give a number indicating the change in pain scores.
  The FLACC (Face, legs, activity, cry and consolability) Scale, ranging from 0 (no pain) to 10 (worst pain), was used to assess pain.
Time Frame: 3 min
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | J Tip Noise | Pain Ease | J Tip
Number analyzed (Participants) | 56 | 53 | 96
units on a scale | 1.71 (0.42) | 2.82 (0.45) | 0.23 (0.28)
Statistical Analysis 1: Comparison: J Tip Noise vs Pain Ease vs J Tip; Test type: Superiority or Other; p = 0.0001, Kruskal-Wallis

5. Secondary Outcome: Pain at J-tip Deployment
Description: Pain when J-tip deployed assessed by video reviewers using pain scale. The FLACC (Face, legs, activity, cry and consolability) Scale, ranging from 0 (no pain) to 10 (worst pain), was used to assess pain.
Time Frame: 1 minute
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | J Tip Noise | Pain Ease | J Tip
Number analyzed (Participants) | 56 | 53 | 96
units on a scale | 3.25 [0.5 to 7.25] | 2.5 [0.5 to 6.5] | 4.0 [0.5 to 8.5]
Statistical Analysis 1: Comparison: J Tip Noise vs Pain Ease vs J Tip; Test type: Superiority or Other; p = 0.37, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Patients were assessed for serious events immediately following venipuncture and then the next day via phone follow up.
Description: All patients were assessed for serious adverse events in the lab. Attempts were made to contact the families of all patients the next day for follow up. The research team was unable to contact some families for follow up, therefore the number of patients assessed for Other Adverse Events is smaller than those assessed for Serious Adverse Events.
Arm/Group | J Tip Noise | Pain Ease | J Tip
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/53 | 0/96
Other Adverse Events (participants affected / at risk) | 6/46 | 6/46 | 13/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | J Tip Noise (N=46) | Pain Ease (N=46) | J Tip (N=83)
Bruise present at 24 hours (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 12 (12)
Redness (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Other/Not Specified (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No